CLINICAL TRIAL: NCT05182814
Title: Efficacy Testing of Collagen Drink on Skin Beauty and Sleep Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 21-102-B
Record Dates: First submitted 2022-01-04; First posted 2022-01-10 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-03

CONDITIONS: Skin Condition; Sleep Disturbance
MeSH Terms: conditions — Skin Diseases; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo drink
- Collagen drink (Experimental)
  Interventions: Dietary Supplement: Collagen Juice Drink

INTERVENTIONS:
Dietary Supplement: Placebo drink — Blank
  Arms: Placebo drink
Dietary Supplement: Collagen Juice Drink — Testing product
  Other Names: LISAVEI® Collagen Juice Drink
  Arms: Collagen drink

SUMMARY:
To assess Collagen Drink on skin condition and sleep quality improvement

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged above 20 years old

Exclusion Criteria:

* Subject who is not willing to participate in this study.
* Patients with diseases of the skin, liver, kidney.
* Subjects who have known cosmetic, drug or food allergies, difficulty in digestive tract absorption or disorder.
* Female who is pregnant or nursing
* Constant drug use
* Received facial laser therapy, chemical peeling or UV overexposure (>3 hours everyday) in the past 4 weeks.
* Students taught by the PI

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
The change of skin wrinkles | Change from Baseline skin wrinkles at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin wrinkles. Units: arbitrary units
The change of skin texture | Change from Baseline skin texture at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin texture. Units: arbitrary units
The change of skin collagen density | Change from Baseline skin collagen density at 8 weeks
  DermaLab® Series SkinLab Combo was utilized to measure skin pores. Units: arbitrary units
The change of skin elasticity | Change from Baseline skin elasticity at 8 weeks
  Cutometer® MPA580 was utilized to measure skin elasticity. Units: arbitrary units
The change of skin L* value | Change from Baseline L* value at 8 weeks
  Chroma Meter MM500 was utilized to measure skin L* value. Units: arbitrary units, 0-100
The change of sleep quality | Change from Baseline sleep quality at 8 weeks
  Self-assessment questionnaire was utilized to survey sleep quality.
The change of AGEs of blood | Change from Baseline AGEs at 8 weeks
  Venous blood was sampled to measure AGEs
The change of TIMP-1 of blood | Change from Baseline TIMP-1 at 8 weeks
  Venous blood was sampled to measure TIMP-1
The change of desmosine of blood | Change from Baseline desmosine at 8 weeks
  Venous blood was sampled to measure desmosine

SECONDARY OUTCOMES:
The change of skin melanin index | Change from Baseline skin melanin index at 8 weeks
  Soft Plus was utilized to measure skin melanin index. Units: arbitrary units
The change of skin pores | Change from Baseline skin pores at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin pores. Units: arbitrary units
The change of skin a* value | Change from Baseline skin a* value at 8 weeks
  Chroma Meter MM500 was utilized to measure skin a* value. Units: arbitrary units
The change of skin hydration | Change from Baseline skin hydration at 8 weeks
  Corneometer® CM825 was utilized to measure skin hydration. Units: arbitrary Corneometer® units 0-120
The change of transepidermal water loss | Change from Baseline transepidermal water loss at 8 weeks
  Tewameter® TM300 was utilized to measure skin hydration. Units: g/hm²

CONTACTS AND LOCATIONS:
Locations (1):
- Chia Nan University of Pharmacy ＆ Science, Tainan, Taiwan